CLINICAL TRIAL: NCT05563233
Title: The Effect of ShotBloker and Helfer Skin Tap Technique on Pain and Fear During Intramuscular Injection in Children Aged 6-12 in the Pediatric Emergency Unit
Brief Title: ShotBloker and Helfer Skin Tap Technique During Intramuscular Injection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1824
Record Dates: First submitted 2022-09-06; First posted 2022-10-03 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Pain, Acute; Fear; Emergencies; Child, Only; Injection Fear
MeSH Terms: conditions — Acute Pain; Emergencies; Iatrophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Helfer Skin Tap (Experimental): Helfer Skin Tap (rhythmic tapping of the skin at the injection site to relax the muscles during injection) is an effective method in reducing pain in intramuscular applications in studies performed with the injection technique.
  Before the injection, the observer nurse will fill in the demographic data form, measure the child's heart rate, blood pressure and SpO2 values, and apply the pain and fear assessment scale. In addition, the pain and fear scale will be evaluated by the child and the parent.
  During the intramuscular injection to be applied to the ventrogluteal region, the level of pain and fear will be examined using the Helfer skin tap technique.
  5 minutes after the injection, the pain and fear level of the children in all groups will be re-evaluated by the child, the mother and the observing nurse. After the procedure, pulse, blood pressure and SpO2 values will be measured and recorded by the observing nurse.
  Interventions: Other: Helfer skin tap technique
- Shotblocker (Experimental): Shotblocker is a flat, horseshoe-shaped device with short, non-sharp 2 mm thick blunt protrusions that connect with the skin, and a hole in the middle to expose the injection site used to reduce pain during subcutaneous or intramuscular injection applications.
  Before the injection, the observer nurse will fill in the demographic data form, measure the child's heart rate, blood pressure and SpO2 values, and apply the pain and fear assessment scale. In addition, the pain and fear scale will be evaluated by the child and the parent.
  During the intramuscular injection to be applied to the ventrogluteal region, the level of pain and fear will be examined by using Shot Blocker.
  5 minutes after the injection, the pain and fear levels of the children in all groups will be re-evaluated by the child, the mother and the observing nurse. After the procedure, pulse, blood pressure and SpO2 values will be measured and recorded by the observing nurse.
  Interventions: Device: Shot Blocker
- control group (No Intervention): Before the injection, the observer nurse will fill in the demographic data form, measure the child's heart rate, blood pressure and SpO2 values, and apply the pain and fear assessment scale. In addition, the pain and fear scale will be evaluated by the child and the parent.
  The level of pain and fear will be examined during intramuscular injection into the ventrogluteal region without any intervention.
  5 minutes after the injection, the pain and fear level of the children in all groups will be re-evaluated by the child, the mother and the observing nurse. After the procedure, pulse, blood pressure and SpO2 values will be measured and recorded by the observing nurse.

INTERVENTIONS:
Other: Helfer skin tap technique — Using the Helfer skin tap technique during intramuscular injection to the ventrogluteal region.
  Arms: Helfer Skin Tap
Device: Shot Blocker — Shot Blocker will be used during intramuscular injection to be applied to the ventrogluteal region.
  Arms: Shotblocker

SUMMARY:
To examine the effect of the Helfer skin tap technique and ShotBloker application on pain and fear experienced during intramuscular injection in children aged 6-12 in the pediatric emergency unit. It was planned as a randomized controlled experimental study to determine its effect on fear. The population of the study will be children aged 6-12 years who applied to the Tarsus State Hospital, and Pediatric Emergency Clinic and the sample will be 177 children who will undergo intramuscular intervention and meet the criteria for inclusion in the study. In data collection; Data collection form, Wong-Baker Scale, and Child fear scale will be used. In order to examine the mean scores of pain and fear according to intramuscular administration techniques in children, appropriate tests will be used by making an analysis of conformity to normal distribution.

DETAILED DESCRIPTION:
Pain is an experience of complex perceptions that overwhelms the patient, distorts their behavior and thoughts, prompts them to perform activities that require immediate attention and aim to stop the pain, and causes behavioral reactions and automatic changes.

To examine the effect of the Helfer skin tap technique and ShotBloker application on pain and fear experienced during intramuscular injection in children aged 6-12 in the pediatric emergency unit.

Type of Study: It was planned as a randomized controlled experimental study to determine the effect of Helfer skin tap technique and Shot Blocker application on pain and fear experienced during intramuscular injection in children aged 6-12 years who applied to the pediatric emergency clinic.

Research Population and Sample Selection The population of the study will be children aged 6-12 years who applied to the Tarsus State Hospital, Pediatric Emergency Clinic, and the sample will be 177 children who will undergo intramuscular intervention, meeting the criteria for inclusion in the research. According to the results of the G-power analysis for the sample size, in accordance with the literature of Canbulat and Bal (2015), Canbulat et al (2014) and Mutlu (2012) to find a medium power effect size difference of 0.25 between the groups, type I error 0.05, power of the test. While 0.80 (α= 0.05, β= 0.20), the minimal sample size was 177 (n=59 for each group).

Data collection Stages of Research Stage 1: A pilot study will be conducted with 20 children in order to evaluate the appropriateness of the forms and scales used before the research.

Stage 2: The purpose of the research and how to record the data will be explained to the nurse who will administer the intramuscular injection procedure using the ventrogluoteal region and to the nurse who will observe the child's pain and fear during the procedure. The children in the sample group and their parents will be informed about the path followed in practice and the research, and their verbal and written consent will be obtained.

Stage 3: The patients who meet the sample selection criteria will be randomly and equally distributed into 3 groups through a program in the computer environment, and randomization will be provided.

(http://www1.assumption.edu/users/avadum/applets/RandAssign/GroupGen.html) (1st experimental group Helfer skin tap technique suitable group, 2nd experimental group Shot Blocker group, 3rd group control group) Children in each group will be provided with their parents.

Stage 4: The nurse observing the children in all groups before the procedure will fill in the demographic data form, measure the child's pulse, blood pressure and SpO2 values, and apply the pain and fear assessment scale. In addition, the pain and fear scale will be evaluated by the child and the parent.

Stage 5: Intramuscular injection will be given to the ventrogluoteal region by following the procedure steps for the children in all groups. The intramuscular injection procedure will be performed by the same nurse. During the procedure, the child's pain and fear will be observed by the observing nurse and recorded in the observation form.

At this stage;

* First Experimental group; During the intramuscular injection to be applied to the ventrogluoteal region, the level of pain and fear will be examined using the Helfer skin tap technique.
* Second Experiment group; During the intramuscular injection to be applied to the ventrogluoteal region, the level of pain and fear will be examined by using Shot Blocker.
* To the control group; The level of pain and fear will be examined during intramuscular injection into the ventrogluotealregion without any intervention.

Stage 6: 5 minutes after the procedure, the pain and fear level of the children in all groups will be re-evaluated by the child, the mother and the observing nurse. After the procedure, pulse, blood pressure and SpO2 values will be measured and recorded by the observing nurse.

Stage 7: The analysis and reporting of the obtained data will be done.

ELIGIBILITY:
Inclusion Criteria:

* To be 6-12 years old,
* Volunteering to participate in the research,
* Not having a chronic disease, not having a mental or neurological disability,
* Being able to communicate verbally,
* Not taking any medication that has an analgesic effect at least 6 hours before applying to the emergency room.
* Not have a life-threatening (sepsis, shock, respiratory/cardiogenic arrest, etc.) disease

Exclusion Criteria:

* Not to be between the ages of 6-12,
* Not volunteering to participate in the research,
* Having a chronic disease, mental or neurological disability,
* Taking any analgesic medication at least 6 hours before applying to the emergency room
* Having a life-threatening (sepsis, shock, respiratory/cardiogenic arrest, etc.) disease

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Scale score | 1 day
  Wong-Baker Scale (Pain Face Rating Scale): In the Wong-Baker scale, there are faces representing increasing pain severity from left to right, ranging from zero to five. The leftmost face has a smiling expression, indicating a pain-free state, while the right-most face has a crying expression, corresponding to the most severe pain. Below each facial expression is a short description describing the severity of pain: 0 - no pain, 1- a little pain, 2- a little more pain, 3- even more pain, 4- a lot of pain, 5- the most severe pain.
  Before, during, and 5 minutes after the injection, the pain level of the children in all groups will be re-evaluated.
Child Fear Scale score | 1 day
  Child Fear Scale: The Child Fear Scale is a scale used to assess the anxiety level of children with 5 face shapes scored between 0-4. 0 = no anxiety, 4 = severe anxiety.
  Before, during, and 5 minutes after the injection, the fear level of the children in all groups will be re-evaluated.
mean arterial pressure | 1 day
  The mean arterial pressureof the child was evaluated and recorded before during, and 5 minutes after the injection
heart rate | 1 day
  The heart rate of the child was evaluated and recorded before during, and 5 minutes after the injection
saturation | 1 day
  The saturation of the child was evaluated and recorded before during, and 5 minutes after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Sönmez Düzkaya, Principal Investigator — Tarsus University; Senem Andı, Principal Investigator — Tarsus Univesity
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin E, Avsar G. Examining the effect of "Shotblocker" in relieving pain associated with intramuscular injection. Complement Ther Med. 2019 Dec;47:102192. doi: 10.1016/j.ctim.2019.09.001. Epub 2019 Sep 3. PMID 31779992
- [Background] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- [Background] Aykanat Girgin, B., Aktaş E., Kılınç, D., Gözen, D. (2020). Let's Prefer the Pain Reducing Intervention, Buzzy or ShotBlocker: A Randomized Controlled Trial. Journal of Behçet Uz Children's Hospital, 10(3),290-298.
- [Background] Bilge S, Aydin A, Gun C, Aldinc H, Acar YA, Yaylaci S, Cinar O, Balci V. Comparison of the efficacy of ShotBlocker and cold spray in reducing intramuscular injection-related pain in adults. A prospective, randomized, controlled trial. Saudi Med J. 2019 Oct;40(10):996-1002. doi: 10.15537/smj.2019.10.24322. PMID 31588477
- [Background] Sivri Bilgen B, Balci S. The Effect on Pain of Buzzy(R) and ShotBlocker(R) during the Administration of Intramuscular Injections to Children: A Randomized Controlled Trial. J Korean Acad Nurs. 2019 Aug;49(4):486-494. doi: 10.4040/jkan.2019.49.4.486. PMID 31477677
- [Background] Canbulat Sahiner N, Turkmen AS, Acikgoz A, Simsek E, Kirel B. Effectiveness of Two Different Methods for Pain Reduction During Insulin Injection in Children With Type 1 Diabetes: Buzzy and ShotBlocker. Worldviews Evid Based Nurs. 2018 Dec;15(6):464-470. doi: 10.1111/wvn.12325. Epub 2018 Oct 11. PMID 30307692
- [Background] Celik N, Khorshid L. The Use of ShotBlocker for Reducing the Pain and Anxiety Associated With Intramuscular Injection: A Randomized, Placebo Controlled Study. Holist Nurs Pract. 2015 Sep-Oct;29(5):261-71. doi: 10.1097/HNP.0000000000000105. PMID 26263287
- [Background] Cobb JE, Cohen LL. A randomized controlled trial of the ShotBlocker for children's immunization distress. Clin J Pain. 2009 Nov-Dec;25(9):790-6. doi: 10.1097/AJP.0b013e3181af1324. PMID 19851160
- [Background] Emel, T., Nese, C., & Leyla, K. (2017). Effects of ShotBlocker on relief of pain due to Hepatitis B vaccine injection into deltoid muscle. International Journal of Caring Sciences, 10(3), 1669-75
- [Background] Jose, R. M., Sulochana, B., & Shetty, S. (2012). Effectiveness of Skin Tap Technique in Reducing Pain Response. International Journal of Nursing Education, 4(1).
- [Background] Khanra, S., & Lenka, A. (2018). Helfer Skin Tap Technique on Pain Associated With Intramuscular Injection among Adult Patients. International Journal of Nursing Education, 10(3), 12-17.
- [Background] Mahato, E. (2019). Effectiveness of Helfer's Skin Tap Technique Versus Routine Technique on Pain Reduction among Patients Receiving Intramuscular Injections. International Journal of Nursing Education, 11(1),41-44.
- [Background] Serena S. Rhythmic skin tapping: an effective measure to reduce procedural pain during IM injection. Nurs J India. 2010 Aug;101(8):178-80. No abstract available. PMID 23520823
- [Background] Soliman, H. M. M., & Hassnein, A. A. (2016). Efficacy of Helfer skin tapping technique on pain intensity as perceived by the patients receiving intramuscular injection. International Journal of Nursing Didactics, 6(2), 12-22.
- [Background] Therese, A. M., & Devi, S. (2014). Effectiveness of Helfer skin tap technique and . routine technique on pain reduction among patients receiving intramuscular injection at Government General Hospital, Puducherry. Int J Sci Res, 3(10).
- [Background] Yilmaz G, Alemdar DK. Using Buzzy, Shotblocker, and Bubble Blowing in a Pediatric Emergency Department to Reduce the Pain and Fear Caused by Intramuscular Injection: A Randomized Controlled Trial. J Emerg Nurs. 2019 Sep;45(5):502-511. doi: 10.1016/j.jen.2019.04.003. Epub 2019 Jun 27. PMID 31257044